CLINICAL TRIAL: NCT04265547
Title: Family-Based Intervention Study of the Effects of Environmental Exposures on Breast Tissue Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); National Cancer Institute (NCI) (NIH); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Mary B. Terry, Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAS2359; 5U01ES026127-04 (NIH)
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Risk
Keywords: Breast Cancer; Xenoestrogen; Household Intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Mother-daughter pairs will partake in an educational session at the baseline visit, which will cover topics on reading product labels, cleaning habit, and cooking methods for reducing environmental exposures. Educational materials will be adapted from the Environmental Protection Agency (EPA) and other accredited sources. Participants will also be introduced to free resources for consumer product safety information, such as the Detox Me phone application. Participants in the intervention arm will receive a 6-month supply of soap, lotion, deodorant, lip balm, a mop, cleaning cloths, and an air filter to take home with them. Mother-daughter pairs in both study arms will return for a second clinic visit 6 months after the pre-intervention visit for blood and urine sample collection, Optical Spectroscopy (OS) measurement, and questionnaire completion.
  Interventions: Behavioral: Breast Cancer Risk Reduction Household Intervention
- Control Arm (No Intervention): Mother-daughter pairs will partake in an educational session at the baseline visit, which will cover topics on reading product labels, cleaning habit, and cooking methods for reducing environmental exposures. Educational materials will be adapted from the Environmental Protection Agency (EPA) and other accredited sources. Participants will also be introduced to free resources for consumer product safety information, such as the Detox Me phone application. Mother-daughter pairs in both study arms will return for a second clinic visit 6 months after the pre-intervention visit for blood and urine sample collection, Optical Spectroscopy (OS) measurement, and questionnaire completion. Control arm participants will be offered the chemical-free products, cleaning supplies, and air filter at this time.

INTERVENTIONS:
Behavioral: Breast Cancer Risk Reduction Household Intervention — This study will focus the intervention on ways at the individual level to reduce sources of Polycyclic Aromatic Hydrocarbons (through cooking methods, exposure to cigarette smoking, indoor air filters) and also individual ways to reduce sources of other Endocrine Disrupting Chemicals. Mother-daughter pairs will partake in an educational session at the baseline visit, covering topics on reading labels, cleaning habits, and cooking methods for reducing exposures. Participants will also be introduced to free resources for consumer product safety information. The intervention arm will receive a 6-month supply of soap, lotion, deodorant, lip balm, a mop, cleaning cloths, and an air filter to take home with them. Pairs in both study arms will return for a second clinic visit 6 months after the pre-intervention visit for blood and urine sample collection, Optical Spectroscopy measurement, and questionnaire completion. The control arm will be offered the intervention products at this time.
  Arms: Intervention Arm

SUMMARY:
This research study is being conducted to find out whether changes in household and personal behavior aimed at reducing exposure to environmental chemicals in dust (increased house dust removal efforts/cleaning and hand washing) and consumer products (increased us of personal care and beauty products that are free of chemicals including phthalates, parabens, and phenols) results in lower exposure to environmental chemicals including polycyclic aromatic hydrocarbons (PAHs) and endocrine disrupting chemicals including phthalates, parabens and phenols. These chemicals may have harmful health effects, as they can interfere with normal functions of the body. This study will also assess changes in breast tissue composition to understand the role of environmental exposures in breast cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* Participant of Columbia's Breast Cancer Research and the Environment (BCERP) Study that recruited from the Columbia Children's Center for Environmental Health (CCCEH) Mothers and Newborns cohort.
* Mother did not smoke or use illicit drugs prior to or during pregnancy (referring to pregnancy for participating daughter).
* Mother was 18-35 years at time of daughter's delivery.
* Mother registered in the prenatal clinics by the 20th week of pregnancy.
* Mother free of diabetes, hypertension and reported HIV infection.
* Mother resided in northern Manhattan or the South Bronx neighborhoods of New York City for at least one year prior to pregnancy.
* Mother self-identified as African-American or Dominican.
* Only participants in the CCCEH birth cohort who answered in the affirmative to the question "I would like to be contacted about future studies" on the consent form of the Mothers and Newborns Study will be contacted to participate in this intervention.

Exclusion Criteria:

• None

Ages: 10 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of measuring pre/post-intervention change in participants' breast tissue concentration of lipid (mg/cm^3) measured using an Optical Spectroscopy machine. | Baseline, 6 months
  Breast tissue composition will be assessed at each clinic visit using an Optical Breast Spectroscopy machine, a minimally invasive procedure that is investigational and not currently FDA-approved. This machine places a light source on 4 different locations of the breast (at 12, 3, 6, and 9 o'clock) and reads the reflected light through the breast tissue. The OS exam will be completed twice on each side of the chest so that 8 measures are taken from the left breast and 8 measures will be taken from the right breast (with each measurement taking no more than a minute). A Monte-Carlo light propagation simulation technique (FullMonte) will be used to extract breast tissue concentration of lipid (mg/cm^3).
Feasibility of measuring pre/post-intervention change in participants' breast tissue concentration of water (mg/cm^3) measured using an Optical Spectroscopy machine. | Baseline, 6 months
  Breast tissue composition will be assessed at each clinic visit using an Optical Breast Spectroscopy machine, a minimally invasive procedure that is investigational and not currently FDA-approved. This machine places a light source on 4 different locations of the breast (at 12, 3, 6, and 9 o'clock) and reads the reflected light through the breast tissue. The OS exam will be completed twice on each side of the chest so that 8 measures are taken from the left breast and 8 measures will be taken from the right breast (with each measurement taking no more than a minute). A Monte-Carlo light propagation simulation technique (FullMonte) will be used to extract breast tissue concentration of water (mg/cm^3).
Feasibility of measuring pre/post-intervention change in participants' breast tissue concentration of collagen (mg/cm^3) measured using an Optical Spectroscopy machine. | Baseline, 6 months
  Breast tissue composition will be assessed at each clinic visit using an Optical Breast Spectroscopy machine, a minimally invasive procedure that is investigational and not currently FDA-approved. This machine places a light source on 4 different locations of the breast (at 12, 3, 6, and 9 o'clock) and reads the reflected light through the breast tissue. The OS exam will be completed twice on each side of the chest so that 8 measures are taken from the left breast and 8 measures will be taken from the right breast (with each measurement taking no more than a minute). A Monte-Carlo light propagation simulation technique (FullMonte) will be used to extract breast tissue concentration of collagen (mg/cm^3).
Feasibility of measuring pre/post-intervention change in participants' breast tissue concentration of total hemoglobin (μM) measured using an Optical Spectroscopy machine. | Baseline, 6 months
  Breast tissue composition will be assessed at each clinic visit using an Optical Breast Spectroscopy machine, a minimally invasive procedure that is investigational and not currently FDA-approved. This machine places a light source on 4 different locations of the breast (at 12, 3, 6, and 9 o'clock) and reads the reflected light through the breast tissue. The OS exam will be completed twice on each side of the chest so that 8 measures are taken from the left breast and 8 measures will be taken from the right breast (with each measurement taking no more than a minute). A Monte-Carlo light propagation simulation technique (FullMonte) will be used to extract breast tissue concentration of total hemoglobin (μM).
Feasibility of measuring pre/post-intervention change in participants' breast tissue concentration of oxygenated hemoglobin (%) measured using an Optical Spectroscopy machine. | Baseline, 6 months
  Breast tissue composition will be assessed at each clinic visit using an Optical Breast Spectroscopy machine, a minimally invasive procedure that is investigational and not currently FDA-approved. This machine places a light source on 4 different locations of the breast (at 12, 3, 6, and 9 o'clock) and reads the reflected light through the breast tissue. The OS exam will be completed twice on each side of the chest so that 8 measures are taken from the left breast and 8 measures will be taken from the right breast (with each measurement taking no more than a minute). A Monte-Carlo light propagation simulation technique (FullMonte) will be used to extract breast tissue concentration of oxygenated hemoglobin (%).
Feasibility of measuring pre/post-intervention change in urinary metabolites of endocrine disrupting chemicals, including polycyclic aromatic hydrocarbons (PAH), phthalates, and parabens (all measured in μg/L units) . | Baseline, 6 months
  Spot urines will be collected from mothers and daughters in each study arm at the pre-intervention and post-intervention clinic visits. Samples will be processed, aliquoted, and stored at -80°C within two hours of collection. Urinary concentrations of metabolites (μg/L) of PAH, phthalates and parabens will be measured in urine samples using commercially available ELISA kits. Blood samples will also be collected at pre- and post-intervention clinic visits using standard protocol, with the buffy coat of white blood cells, packed red blood cells, and plasma separated and stored in multiple aliquots at -80°C for future analyses. Each urine and blood sample will receive a unique barcode, blinding the lab technician to the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Terry, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Mailman School of Public Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No